CLINICAL TRIAL: NCT01998763
Title: Knowledge Innovation Project of CAS - Genetic and Nutritional Association Studies on Metabolism-related Diseases in Chinese Population -- Vitamin D Intervention Study
Brief Title: Vitamin D Intervention Trial in Healthy Chinese, Phase II
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Xu Lin, Principal Investigator, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KSCX2-EW-R-10-VDII; KSCX2-EW-R-10 (Other Grant/Funding Number: Knowledge Innovation Project of CAS)
Record Dates: First submitted 2013-11-25; First posted 2013-12-02 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D3 supplementation; metabolite profile; SNPs; bone-turnover marker
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 5 placebo pills per day, 20 weeks
  Interventions: Dietary Supplement: Placebo
- 2000 IU/d Vitamin D3 (Experimental): 5 vitamin D3 pills per day, 20 weeks
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Placebo — placebo capsules have similar appearance and smell as 400 IU vitamin D3 capsules,
  Arms: Placebo
Dietary Supplement: Vitamin D3 — Vitamin D3 2000 IU per day
  Arms: 2000 IU/d Vitamin D3

SUMMARY:
This is a double-blind, randomized, placebo-controlled trial. Based on inclusion and exclusion criteria, 400 eligible volunteers, who were 20-45 years, with 25-hydroxyvitamin D between 12.5-50 nmol/L and BMI between 18.5-28 kg/m2, were enrolled and randomly assigned to placebo or 2000 IU/d vitamin D3 arm, after taking placebo for one week. The study protocol was approved by the Ethics Committee of Huadong Hospital Affiliated to Fudan University, Shanghai and all participants provided written informed consents.In this 2-arm RCT we aimed to systematically investigate the effect of:

1. vitamin D3 supplement on serum 25(OH)D levels and the modifying factors;
2. genetic and non-genetic variants on vitamin D bioavailability;
3. vitamin D3 supplementation on metabolic profiles and circulating bone-turnover markers

DETAILED DESCRIPTION:
At present time, the Recommended Dietary Allowance (RDA) and the tolerable upper intake level (UL) for vitamin D are 200 IU/day and 800 IU/day for Chinese aged 11-50 years, respectively. On the other hand, the RDA and UL for vitamin D for the same age group in USA are 600IU/day and 4000IU/day, respectively. Indeed, recent epidemiological studies suggested that serum 25-hydroxyvitamin D [25(OH)D] concentration ≥75 nmol/L appeared to be optimal for preventing cardiometabolic diseases and improving bone health. To achieve this goal, a daily intake of 1000 IU or equivalent amount from other sources, is needed, which is twice as much as the RDA recommended by Chinese Nutrition Society. Except for those individuals with hypersensitive conditions, daily intake less than 10,000 IU of vitamin D have not shown overt adverse effects based upon the studies conducted in Western populations.

Since vitamin D metabolic rate and its relationship with health outcomes may vary across different ethnical groups and most available data so far were from Caucasians populations, it remains to be elucidated whether the findings from Western population could apply directly to Asian peoples like Chinese. Recently, our group has conducted the first relatively large-scale study in Asian to evaluate the association between 25(OH)D and risk of metabolic syndrome. It was found that the geometric mean of plasma 25(OH)D in these Chinese adults aged 50-70 years from Beijing and Shanghai (n=3210) was 40.36 nmol/l and percentage of vitamin D deficiency [25(OH)D <50 nmol/l] and insufficiency (50 ≤ 25(OH)D < 75 nmol/l) were 69.2% and 24.4%, respectively. Comparing the lowest with the highest 25(OH)D quintile (≤28.7 nmol/l vs. ≥57.7 nmol/l), the odds ratio for metabolic syndrome (MetS) was 1.52 (95% CI 1.17-1.98, P for trend = 0.0002), after multiple adjustment. Significant inverse associations also existed between 25(OH)D and most of MetS components, plus HbA1c. Moreover, low plasma 25(OH)D level was found to be associated with increased insulin resistance index (homeostasis model assessment of insulin resistance, HOMA-IR) in those overweight and obese individuals (BMI ≥24 kg/m2),. (Lu et al., Diabetes Care, 2009). According to the data from 2002 China National Nutrition Survey, high prevalence of vitamin D deficiency also exited in Chinese children aged 1-3 years and approximate 82% of them had circulating 25(OH)D ≤ 50nmol/L. In consistent with our finding, a report from a population-based Korea study showed that the association between 25(OH)D and insulin resistance was modified by BMI status (Choi et al.,The Journal of Nutrition,2011).

In our recent genetic study, it was found that genetic variants at GC and NADSYN1/DHCR7 were significantly associated with circulating 25(OH)D levels while marginal association between CYP2R1-rs2060793 and 25(OH)D levels was observed only in the Shanghai subpopulation (Lu et al., Human Genetics 2011). In addition, we developed a genetic risk score (GRS) to evaluate the combined effect of three SNPs (rs4588, rs1790349 and rs2060793) from GC, NADSYN1/DHCR7 and CYP2R. Notably, the average plasma 25(OH)D concentration in individuals with 5-6 risk allele was 11.4 nmol/l lower than those without risk allele. Indeed, previous studies suggested that intake of 100 IU vitamin D could only raise circulating 25(OH)D by 2.5 nmol/l, implicating that 450 IU of extra vitamin D is required for these high risk individuals. The possible interpretations for such a high prevalence of poor vitamin D nutrition among Chinese may be due to the factors: (1) unlike United States and other Western countries, few, if any, vitamin D enriched or fortiﬁed foods are available in China; (2) Chinese, particularly women, like to have pale skin color, who therefore frequently utilize sunscreen and umbrella to prevent sun exposure. (3) approximate 318 million people are living in Heilongjiang, Shaanxi, Jilin, Shanxi, Liaoning, Qinghai, Gansu, Inner Mongolia, Xinjiang, and Hebei provinces, the areas with latitude N37°, which was previously showed to prevent skin synthesizing sufficient vitamin D during winter time. Collectively, all of these factors suggest that large proportions of Chinese may suffer vitamin D insufficiency or deficiency whereas the current RDA in China might be too low to provide adequate vitamin D for people's health. In order to fill up this gap, therefore, it is essential to study the bioavailability following vitamin D intervention and also identify the effects of genetic variants and other factors on vitamin D metabolism and associated health outcomes. Ultimately, the current study will provide important evidence for establishing optimal vitamin D requirement for Chinese people.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-45 years. with vitamin D deficiency (12.5 ≤ 25(OH)D < 50 nmol/l)

Exclusion Criteria:

* BMI < 18.5 kg/m2, or BMI ≥ 25 kg/m2
* Total intake of calcium from diet or supplements >1200mg/d, or fasting serum calcium level ≥2.75 mmol/l
* Participating in other clinical studies within previous 3 months
* Taking vitamin D supplements within previous 3 months
* Using medications that may affect vitamin D metabolism in previous 3 months;
* Concomitant with clinical conditions, like liver dysfunction (serum alanine transaminase (ALT) ≥40 U/L; and/or aspartate transaminase (AST) ≥40 U/L; Glutamyl transpeptidase （GGT）≥50 U/L; serum creatinine < 50 or > 120 µmol/L; urea nitrogen (UN) < 7 or > 18 mg/dl, and/or urine acid <90 or >420 µmol/L; which may affect vitamin D metabolism;
* History of drug or alcohol abuse (>40 g/d)
* Women during pregnancy or lactation
* Individuals with mental disorders or current use of antidepressants, the conditions which may affect him or her understanding and unwillingness to the intervention;
* Having clinically diagnosed AIDS, hepatitis A, hepatitis B, tuberculosis and other infectious diseases.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 448 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
25-hydroxyvitamin D | 0,10,20 week
  Serum 25(OH)D (D2+D3) concentration was measured by a liquid chromatography-mass spectrometry (LC-MS) method

SECONDARY OUTCOMES:
calcium | 0,10,20 week
  Serum calcium was measured by an automatic biochemical analyzer
parathyroid hormone | 0,10,20 week
  Serum iPTH was measured by ADVIA Centaur XP Immunoassay System (Siemens, Germany)
Vitamin D binding protein | 0,10,20 week
  Serum VDBP was measured by an ELISA kit

CONTACTS AND LOCATIONS:
Overall Officials: Xu Lin, PhD, Principal Investigator — Institute for Nutritional Sciecnes, Chinese Acadamy of Sciences
Locations (1):
- Institute for Nutritional Sciecnes, Chinese Acadamy of Sciences, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yao P, Sun L, Xiong Q, Xu X, Li H, Lin X. Cholecalciferol Supplementation Promotes Bone Turnover in Chinese Adults with Vitamin D Deficiency. J Nutr. 2018 May 1;148(5):746-751. doi: 10.1093/jn/nxy032. PMID 29897564
- [Derived] Yao P, Sun L, Lu L, Ding H, Chen X, Tang L, Xu X, Liu G, Hu Y, Ma Y, Wang F, Jin Q, Zheng H, Yin H, Zeng R, Chen Y, Hu FB, Li H, Lin X. Effects of Genetic and Nongenetic Factors on Total and Bioavailable 25(OH)D Responses to Vitamin D Supplementation. J Clin Endocrinol Metab. 2017 Jan 1;102(1):100-110. doi: 10.1210/jc.2016-2930. PMID 27768857